CLINICAL TRIAL: NCT01360125
Title: S0106A, Proteomic Signatures Associated With Complete Response (CR) and Complete Continuous Response at One Year (CCR1) Following Cytarabine-Based Induction Chemotherapy in Younger Adult Patients (18-60 Years of Age) With a Newly Diagnosed Non-M3 AML
Brief Title: S0106A, Biomarkers in Samples From Patients With Newly Diagnosed Acute Myeloid Leukemia Treated With Cytarabine-Based Chemotherapy
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S0106A; S0106A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-05-21; First posted 2011-05-25 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia
Keywords: adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — Flow Cytometry

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: proteomic profiling
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer in the laboratory may help doctors predict how well patients will respond to treatment.

PURPOSE: This research study studies biomarkers in samples from patients with newly diagnosed acute myeloid leukemia treated with cytarabine-based chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Training and testing of multiparameter flow cytometry-based cell signaling signature (FC classifier 1) associated with in vivo primary chemoresistance (i.e., non-complete response [NR]) to standard induction therapy in adult patients ≤ 60 years old with a newly diagnosed non-M3 acute myeloid leukemia (AML).
* Training and testing of multiparameter flow cytometry-based cell signaling signature (FC classifier 2) associated with complete continuous response at 1 year (CCR1) in adult patients ≤ 60 years old with a newly diagnosed non-M3 AML who are treated with cytarabine-based induction chemotherapy.
* Identification of signaling signature(s) associated with secondary chemoresistance (i.e., disease relapse) in adult patients ≤ 60 years of age who have longitudinally paired peripheral blood mononuclear cells (PBMC) or bone marrow mononuclear cells (BMMC) samples at diagnosis and at the time of first relapse. (Exploratory)

OUTLINE: Cryopreserved samples are incubated with cytokines (e.g., interleukins), growth factors (e.g., sargramostim [GM-CSF] and filgrastim [G-CSF]), chemotherapeutic agents (e.g., cytarabine, etoposide phosphate), and other modulators. Cells are fixed, permeabilized, and stained with antibodies that recognize extracellular markers in conjunction with intracellular activation-state specific epitopes of designated signaling molecules. Subsequently, cells are analyzed for multiparametric phospho-flow cytometry in a random manner (without knowledge of clinical variables and outcomes) to training and testing sets. Results are then compared with individual patient clinical outcomes.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed non-M3 acute myeloid leukemia (AML)
* Pretreatment and relapsed and/or refractory cryopreserved bone marrow mononuclear cells (BMMCs) and peripheral blood mononuclear cells (PBMCs) available
* Have 2+ vials of pretreatment marrow cells and/or 2+ vials of pretreatment PBMCs in the Southwestern Oncology Group (SWOG) AML/Myelodysplastic Syndrome (MDS) Repository

  * Usable samples must contain approximately 1.6 ×10^6 cluster of differentiation antigen 45+ (CD45+) cells post thaw.
* Eligible and evaluable patients who participated on SWOG-S0106 study

PATIENT CHARACTERISTICS:

* Did not refuse consent for this use of specimens

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients enrolled in S0106 that consented to use of specimens for future reserach
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response to induction chemotherapy (complete response vs non-complete response) (classifier 1) | immediate
CCR1 at 1 year (classifier 2) | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Radich, MD, Principal Investigator — Fred Hutchinson Cancer Center

REFERENCES:
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844